CLINICAL TRIAL: NCT04606615
Title: Skin Barrier Abnormalities and Oxidative Stress Response in the Skin of Atopic Dermatitis Patients With Food Allergy
Brief Title: Skin Barrier Abnormalities and Oxidative Stress Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: ADRN3-CRC
Record Dates: First submitted 2020-10-16; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Atopic Dermatitis; Food Allergy
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Adults: AD + FA: Adults: atopic dermatitis and food allergy to peanut
- Adults: AD - FA: Adults: atopic dermatitis and no food allergy
- Adults: NC: Adults: Normal Control
- Children: AD+ Peanut: Children: atopic dermatitis and food allergy to peanut
- Children: AD + Milk: atopic dermatitis and food allergy to milk
- Children: AD + Egg: atopic dermatitis and food allergy to egg
- Children: AD only: atopic dermatitis and no food allergy
- Children: NC: Normal Control

SUMMARY:
This is a prospective, single-site controlled observational study designed to comprehensively determine whether children and adults with atopic dermatitis (AD) and food allergy (FA) have skin abnormalities which distinguish them from children with AD without FA, and non-atopic (NA) controls.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 1 to 17 years of age inclusive at Screening for the pediatric group, 18-65 years of age for the adult group
2. For all pediatric participants parent guardian must be able to understand and provide informed consent and participant provide assent as applicable per Institutional Review Board (IRB) guidelines and regulations
3. Children: active AD and food allergy to peanut OR active AD and food allergy to milk OR active AD and food allergy to eggs. Adults: active AD and food allergy to peanut. Participant must meet all of the following criteria:

   * Self-report or documentation of a positive oral food challenge to peanut OR egg OR milk or self-report of an allergic reaction to peanut OR egg OR milk within 2 hours of ingestion
   * Skin prick test wheal≥8mm for peanut, milk or egg OR
   * Active AD and no food allergy. Participant must meet all of the following criteria:
   * No personal history or current manifestations of food allergy (based on no self-report of a positive oral food challenge, positive skin test, positive blood test, or allergic reactions)
   * Negative skin prick test (wheal<3mm) to peanut, milk, egg, wheat, soy, shellfish mix, treenuts, and sesame seed OR

NA. Participant must meet all of the following criteria:

* No personal history or current manifestations of AD, asthma, or allergic rhinitis (based on self-report)
* No personal history or current manifestations of food allergy (based on no self-report of a positive oral food challenge, positive skin test, positive blood test, or allergic reactions)
* Negative skin pricktest (wheal<3mm) to peanut, milk, egg, wheat, soy, shellfish mix, treenuts, and sesame seed
* Negative skin prick test(wheal<3mm) to environmental allergens (cat, dog, dustmite, cockroach, and local trees/grasses/weeds/molds)

Exclusion Criteria:

* 1. Inability or unwillingness of a parent guardian (for pediatric participants) to give written informed consent, or participant to give assent, if applicable, or to comply with study protocol 2. Who have any skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous diseases, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease).

  3. Pregnant or lactating females 4. Known or suspected immunosuppression 5. Severe concomitant illness(es) 6. History of serious life-threatening reaction to latex, tape, or adhesives 7. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study 8. Use of biologics within 5 half-lives (if known) or 16 weeks of the Screening Visit 9. Use of an investigational drug within 5 half-lives (if known) or 8 weeks of the Screening Visit 10. Has received immunotherapy within 12 months of the Screening Visit

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will children and adults. We will include children aged 1-17 years. We will enroll up to 20 AD children with food allergy to peanut, up to 20 AD children with food allergy to milk and no peanut allergy, up to 20 AD children with food allergy to eggs and no peanut allergy, up to 20 AD children without a history of food allergy, and up to 20 NA children. In addition, 18-65 old adults will be enrolled, including up to 20 adults with food allergy to peanut, up to 20 adults with AD without history of food allergy and 20 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Transepidermal Water Loss (TEWL) | Day 0
  area under the TEWL curve (AUC) from four non-lesional skin sites assessed. TEWL will be assessed on non-lesional skin prior to tape stripping and repeated after 5, 10, 15, and 20 tape strips.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No